CLINICAL TRIAL: NCT07230626
Title: A Randomized, Open-Label, Controlled, Multicenter Phase 3 Trial of SYS6002 Versus Chemotherapy of Physician's Choice in Recurrent or Metastatic Cervical Cancer After Platinum-containing Chemotherapy and Anti-PD-(L)1 Agent Therapy
Brief Title: SYS6002 vs Chemotherapy in Recurrent or Metastatic Cervical Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS6002-006
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants in this trial will be randomly assigned to one of two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYS6002 (Experimental): SYS6002 monotherapy
  Interventions: Drug: SYS6002
- Chemotherapy (Active Comparator): Investigator's choice of one chemotherapy treatment (topotecan, gemcitabine, pemetrexed, or docetaxel)
  Interventions: Drug: Investigator's Choice of Chemotherapy

INTERVENTIONS:
Drug: SYS6002 — SYS6002，intravenous injection
  Arms: SYS6002
Drug: Investigator's Choice of Chemotherapy — Investigator's choice of chemotherapy means the chemotherapy chosen by investigators/doctors to treat metastatic cervical cancer, including topotecan (1.2 mg/m^2 of by IV on Days 1 to 5, every 21 days), gemcitabine (1000 mg/m^2 by IV on Days 1 and 8, every 21 days), pemetrexed (500 mg/m^2 by IV on Day 1, every 21 days), or docetaxel (75 mg/m^2 by IV on Day 1, every 21 days).
  Arms: Chemotherapy

SUMMARY:
This study is a randomized, open-label, controlled, multicenter phase Ⅲ clinical trial, which aims to evaluate the efficacy and safety of SYS6002 versus investigator's choice of chemotherapy in the treatment of participants with recurrent or metastatic cervical cancer who have failed platinum-containing chemotherapy and PD-1/L1 inhibitor therapy

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 18-75 years (inclusive);
* 2. Histologically confirmed recurrent or metastatic cervical cancer (squamous cell, HPV-associated adenocarcinoma, or adenosquamous), not amenable to resection or chemoradiation with curative intent;
* 3. Subject must have received a platinum-based chemotherapy with anti-PD-(L)1 agent and if was received administered in the adjuvant/neoadjuvant setting subject must have progressed during treatment or within 6 months of treatment completion；received no more than 2 prior systemic therapy in the metastatic/recurrent setting; must have experienced radiographic progression during or after the last treatment regimen;
* 4. An archival tumor tissue sample or a fresh tissue sample should be provided;
* 5. Subjects must have measurable disease according to RECIST (version 1.1);
* 6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* 7. Life expectancy of ≥ 3 months;
* 8. Major organ function meets the relevant laboratory test standards for hematology, renal function, liver function, and coagulation within 7 days prior to treatment;
* 9.Sexually active fertile subjects must agree to use methods of contraception during the study and at least7 months after termination of study therapy and have a negative urine or serum pregnancy test within 7 days prior to randomization;
* 10.Willing to participate in the study, understand the study procedures, and sign a written informed consent form.

Exclusion Criteria:

* 1. Has other histologies not mentioned as part of the inclusion criteria 2;
* 2. Active central nervous system metastases or leptomeningeal metastasis;
* 3. Adverse events from prior antitumor therapy not recovered to ≤ Grade 1 (unless the investigator deems there is no safety risk)；
* 4. Any serious and/or uncontrolled concurrent illness that may interfere with patient's particiation in the study:

  1. Participants with a history of severe cardiovascular disease within 6 months prior to randomization, including but not limited to:

     Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia and third-degree atrioventricular block requiring clinical intervention; corrected QT interval > 480 ms by Fridericia method (Fridericia formula: QTcF = QT/RR^0.33, RR = 60/heart rate); With history of myocardial infarction, unstable angina pectoris, angioplasty and coronary artery bypass surgery; New York Heart Association (NYHA) classification Grade III and above heart failure, and left ventricular ejection fraction (LVEF) < 50% in the tests and examinations during the screening period; Cerebrovascular Accident; Participants with poorly controlled hypertension on medication, with systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg;
  2. Other clinically significant diseases:

HbA1c > 8%; Participants with active keratitis and corneal ulcer, or fundus lesions with a risk of blindness; Grade ≥2 neuropathy prior to randomization; Severe infection within 4 weeks prior to randomization; active infection requiring systemic antibiotics, antiviral, or antifunga therapy within 2 weeks prior to randomization; Active HBV or HCV infection; History of immunodeficiency (HIV-positive, acquired or congenital immunodeficiency, etc.), or organ transplantation; History of another malignancy within 3 years prior to randomization; History of interstitial lung disease (ILD) / non-infectious pneumonia, or current ILD/non-infectious pneumonia, or imaging findings at screening that cannot rule out these condition, except for those who are determined to be risk-free after discussion between the investigator and the sponsor; History of genital tract fistula, except for whose perforations or fistulas that have been treated with resection or repair, and are considered by the investigator to be healed or in remission; Pleural effusion, ascites or pericardial effusion with syptoms or requiring puncture or drainage within 2 weeks prior to randomization;

* 5. Use of other unmarketed clinical investigational drugs or treatments, chemotherapy, radiotherapy targeted therapy within 4 weeks prior to randomization; use of traditional Chinese medicine with anticancer indication, oral fluoropyrimidine drugs, small molecule targeted drug within 2 weeks prior to randomization; use of palliative radiation or local therapy within 2 weeks prior to randomization;with major surgery within 4 weeks prior to randomization;
* 6. Allergy to any component of SYS6002, or humanized monoclonal antibodies;
* 7. Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 3.5 years
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time will be censored at the last date the participant is known to be alive

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3.5 years
  Objective response rate is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) per RECIST v.1.1.
Duration of Response (DOR) | Up to 3.5 years
  DOR is defined as the time from the date of the first confirmed objective response (CR or PR that is subsequently confirmed) to the date of the first documented disease progression (PD) per RECIST v1.1 or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 3.5 years
  The percentage of participants who experience a best response of CR, PR or stable disease (SD).
Progression Free Survival (PFS) | Up to 3.5 years
  PFS is defined as the time from the date of randomization to the first documentation of PD as assessed by investigator per RECIST v.1.1, or death due to any cause, whichever occurs earlier.
Incidence of adverse events | Up to 3.5 years
Incidence of Anti-Drug Antibody (ADA) | Up to 3.5 years
Blood concentration of SYS6002 | Up to 3.5 years